CLINICAL TRIAL: NCT05839015
Title: Efficacy of an Smartphone App Intervention Based on Self-Compassion for Mental Health Among University Students During and After Covid-19: a Randomized Clinical Trial
Brief Title: Efficacy of an Smartphone App Intervention Based on Self-compassion for Mental Health Among University Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Bruno Luis Schaab, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: bruno.schaabUFCSPA
Record Dates: First submitted 2022-10-14; First posted 2023-05-03 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Mental Health Issue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This is group wil use "Eu + Compassivo" app.
  Interventions: Behavioral: mHealth Intervention Based on Self-Compassion
- Control (No Intervention): This group will be made up of a waiting list.

INTERVENTIONS:
Behavioral: mHealth Intervention Based on Self-Compassion — Self-compassion techniques aim at developing compassionate skills for emotion regulation, such as self-kindness, recognition of common humanity, and mindfulness.
  Arms: Intervention

SUMMARY:
Since the beginning of Covid-19, there has been an increase in the incidence of mental disorders and psychopathological symptoms, such as depression, anxiety and stress, among university students. Even with the end of social distancing, many students still have losses in emotional well-being, so psychotherapeutic interventions are important for the recovery and promotion of the mental health of this public. Interventions based on self-compassion have been associated with improving the mental health of different audiences, either by reducing psychopathological symptoms (such as anxiety) or improving positive constructs associated with mental health, such as hope and optimism. One way to administer interventions based on self-compassion is through mHealth technologies, which have been consolidating since the pandemic. Some studies sought to assess the benefits of self-compassion-based interventions administered in the mHealth format among university students suggest that they have acceptability and are effective regarding indicators of emotional well-being. However, in Brazil, there is still no digital intervention for the cultivation of self-compassion among university students, which could help to mitigate the deleterious effects of the pandemic on mental health. Considering this gap, an intervention based on self-compassion administered via a smartphone app called "Eu + Compassivo" was developed. The present study seeks to evaluate its efficacy in mental health indicators, both psychopathological symptoms and Positive Psychology constructs.

ELIGIBILITY:
Inclusion Criteria:

* Must be enrolled in a course that originally works in the face-to-face format
* Having basic knowledge of the use of smartphones
* Owning a smartphone with internet access and the Android or IOS system
* At least mild depressive, anxiety or stress symptoms

Exclusion Criteria

• Diagnosed with any serious and persistent mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Depression | T1 (pre) to T2 (6-week)
  Depression, Anxiety and Stress Scale (DASS-21) - The measure has 21 items arranged in 3 dimensions (depression, anxiety and stress) through a Likert scale ranging from "did not apply to me at all" (0) to "applied to me very much, or most of the time" (3). The sum of the items provides a score between 0 and 21 regarding depression. The higher the score, the greater the depression.
Change in Anxiety | T1 (pre), T2 (6-week)
  Depression, Anxiety and Stress Scale (DASS-21) - The measure has 21 items arranged in 3 dimensions (depression, anxiety and stress) through a Likert scale ranging from "did not apply to me at all" (0) to "applied to me very much, or most of the time" (3). The sum of the items provides a score between 0 and 21 regarding anxiety. The higher the score, the greater the anxiety.
Change in Stress | T1 (pre), T2 (6-week)
  Depression, Anxiety and Stress Scale (DASS-21) - The measure has 21 items arranged in 3 dimensions (depression, anxiety and stress) through a Likert scale ranging from "did not apply to me at all" (0) to "applied to me very much, or most of the time" (3). The sum of the items provides a score between 0 and 21 regarding stress. The higher the score, the greater the stress.
Change in Self-Compassion | T1 (pre), T2 (6-week)
  Self-Compassion Scale - The measure has 26 items scored on a Likert scale, ranging from "almost never" (1) to "almost always" (5). The higher the score, the greater the sel-compassion.
Change in Compassion | T1 (pre), T2 (6-week)
  Santa Clara Brief Compassion Scale - The measure has 5 items arranged on a Likert scale, ranging from "not at all true for me" (1) to "very true for me" (7). The higher the score, the greater the compassion.
Change in Emotional Well-Being | T1 (pre), T2 (6-week)
  Well-being Index (WHO-5) - It is a generic measure that assesses emotional well-being. It has 5 items, ranging from "at no time" (0) to "all the time" (5) on a Likert scale, providing a score that varies between 0 and 25. The higher the score, the greater the emotional well-being.

SECONDARY OUTCOMES:
Change in Hope | T1 (pre), T2 (6-week)
  Adult Dispositional Hope Scale - The instrument has 21 items arranged in a two-dimensional structure (self-centered hope and altruistic hope), scored on a two-column 6-point Likert scale, which express, respectively, the ideas of desire and expectation in relation to the content of each item ( 0 = do not want; 5 = want very much; 0 = do not believe; 5 = believe very much). The higher the score, the greater the hope.
Change in Emotional Self-Regulation | T1 (pre), T2 (6-week)
  Emotional Dysregulation Scale - The measure has 15 items arranged on a 4-point Likert scale, ranging from "none of the times/not at all" (0) to "always" (5). The higher the score, the greater the emotional dysregulation.
Change in Positive Affect | T1 (pre), T2 (6-week)
  The Positive and Negative Affect Schedule (PANAS) - The measure has 20 items arranged on a Likert scale, 10 of which are negative affects and 10 are positive affects, ranging from "very slightly or not at all" (1) to "extremely" (5). The sum of the scores of each item provides a score that varies between 10 and 50 for positive affect. The higher the score, the greater the positive affect.
Change in Negative Affect | T1 (pre), T2 (6-week)
  The Positive and Negative Affect Schedule (PANAS) - The instrument has 20 items arranged on a Likert scale, 10 of which are negative affects and 10 are positive affects, ranging from "very slightly or not at all" (1) to "extremely" (5). The sum of the scores of each item provides a score that varies between 10 and 50 for negative affect. The higher the score, the greater the negative affect.
Change in Optimism | T1 (pre), T2 (6-week)
  Revised Life Orientation Test - The measure has 10 items arranged on a Likert scale ranging from "strongly disagree" (1) to "strongly agree" (5). The higher the score, the greater the optimism.
Change in Life Satisfaction | T1 (pre), T2 (6-week)
  Satisfaction With Life Scale (SWLS) - The measure has 5 items arranged on a Likert scale ranging from "strongly disagree" (1) to "strongly agree" (7). The sum of the scores for each item provides a score between 5 and 35. The higher the score, the greater the life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Tozzi Reppold, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre; Prisla Ücker Calvetti, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre; Sílvio César Cazella, PhD, Principal Investigator — Federal University of Health Sciences of Porto Alegre

IPD SHARING:
Plan to Share IPD: No